CLINICAL TRIAL: NCT00488904
Title: Omega-3 Fatty Acids and Postoperative Complication After Colorectal Surgery
Brief Title: Omega-3 Fatty Acids and Postoperative Complications After Colorectal Surgery
Acronym: omega3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Lone Schmidt Sørensen, Fresenius Kabi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 123omega; VN2005/35
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-04

CONDITIONS: Colorectal Cancer
Keywords: infection; colorectalcancer; omega-3 fedtsyre; complications
MeSH Terms: conditions — Colorectal Neoplasms; Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- a (Experimental)
  Interventions: Dietary Supplement: supportan
- b (Placebo Comparator)
  Interventions: Dietary Supplement: supportan placebo

INTERVENTIONS:
Dietary Supplement: supportan — 2 sip feed pr. day
  Arms: a
Dietary Supplement: supportan placebo — 2 sip feed pr. day
  Arms: b

SUMMARY:
To discover whether an Omega-3 fatty acid (eicosapentaenoic acid/EPA and docosahexaensyre/DHA) enriched nutritional supplement given 7 days preoperatively and 7 days postoperatively may reduce the frequency of postoperative infectious complications defined as: pneumonia, wound infection, urinary tract infection, peritonitis (including anastomotic leakage) and septic conditions of any cause in patients who undergo elective operations for colorectal cancer compared with a nutritional preparation that is identical apart from the EPA content.

DETAILED DESCRIPTION:
Several earlier studies indicate that perioperative supplements of Omega-3 fatty acids can reduce the risk of postoperative complications after major surgery through an immune modulating effect in the form of a downward adjustment of the inflammatory response. (1-7) The interpretation of these studies is made more difficult by differences in their method of administration (parentally/enterally), differences in the time of the intervention (preoperative/postoperative) and differences in the selection of patients (malnourished cancer patients / upper GI cancer patients/mixed surgical patients) and finally because many of the studies deal with a so-called immune modulating preparation containing a mixture of arginine, Omega-3 fatty acids and ribonucleic acid.

The biological effects of fish oils are related to their content of such things as Omega-3 fatty acids that can be incorporated in cell membranes where they influence receptor function, enzyme activity and the production of lipid mediators. The cells from the immune system perform their functions through membrane-associated activities like secretion of cytokines, antibodies, lymphocyte transformation and contact lysine. These functions can be affected by changes in the membrane structure. (7;8) Besides the effect parameter of postoperative septic complications, many of these studies use pseudoparameters such as length of stay, need for respirator treatment, time in intensive care as well as a wide range of biochemical changes whose relevance to the clinic process can be difficult to assess. (1-7;9-13;). It is well-known that early enteral nutrition reduces the risk of postoperative complications (14; 15). Many of the aforementioned studies similarly point to a benefit from using Omega-3 fatty acid enriched nutritional preparations preoperatively. There is now a commercially manufactured nutritional preparation for peroral consumption containing Omega-3 fatty acids - Supportan (Fresenius-Kabi). The preparation is more energy intensive than similar drink preparations, but does not otherwise differ in composition from standard preparations. It is approved by the Danish Veterinary and Food Administration for this study.

In 2 x 200ml of Supportan 3 g EPA and DHA are given daily. In other studies up to 10 g have been given daily without side effects. (6; 16)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients for elective colorectal resection for cancer, ASA group 1-3 (see annex)

Exclusion Criteria:

* Diabetes Mellitus
* Alcohol consumption > 5 drinks per day
* Acute operation
* Non Danish speakers
* Patients with untreated psychiatric conditions
* Pregnant or breast-feeding women
* Patients with ICD-pacemaker
* Patients with reduces kidney function and immunosuppressed patients
* patients that eat or drink omega-3 fatty acids
* patients operated for 2 different cancers in 1 operation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2007-06; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
In previous studies a complication frequency (infectious complications) of at least 30% was found for this type of operation (14; 17) This figure has to be reduced to 10% (MIREDIF = 20%). | 1 year
  Primary outcome measures are infectious complications after surgery for colorectal cancer defined as: pneumonia, cystitis, wound infection, intraabdominal abscess, peritonitis, septicemia, other infections.
  30 day mortality and other complications such as bleeding, wound dehiscence, anastomotic leakage will also be registered

SECONDARY OUTCOMES:
The secondary outcome variable is hospitalisation time and mortality. Given the material's size, it is not expected to be possible to demonstrate a significant reduction in mortality | 1 year
incorporation of fatty acids in cell membranes | after 7 days of intervention
  laboratory test on blood sample (leucocytes
development in interleukins after surgery | day 1-4 after surgery
  analysis of blood sample
lenght of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Erik be schmidt, professor, Study Director — Aalborg Hospital the lipid clinic
Locations (1):
- Aalborg Hospital, Aalborg, Aalborg, Denmark

REFERENCES:
- [Background] Braga M, Gianotti L, Vignali A, Cestari A, Bisagni P, Di Carlo V. Artificial nutrition after major abdominal surgery: impact of route of administration and composition of the diet. Crit Care Med. 1998 Jan;26(1):24-30. doi: 10.1097/00003246-199801000-00012. PMID 9428539
- [Background] Braga M, Gianotti L, Nespoli L, Radaelli G, Di Carlo V. Nutritional approach in malnourished surgical patients: a prospective randomized study. Arch Surg. 2002 Feb;137(2):174-80. doi: 10.1001/archsurg.137.2.174. PMID 11822956
- [Background] Gianotti L, Braga M, Vignali A, Balzano G, Zerbi A, Bisagni P, Di Carlo V. Effect of route of delivery and formulation of postoperative nutritional support in patients undergoing major operations for malignant neoplasms. Arch Surg. 1997 Nov;132(11):1222-9; discussion 1229-30. doi: 10.1001/archsurg.1997.01430350072012. PMID 9366716
- [Background] Schilling J, Vranjes N, Fierz W, Joller H, Gyurech D, Ludwig E, Marathias K, Geroulanos S. Clinical outcome and immunology of postoperative arginine, omega-3 fatty acids, and nucleotide-enriched enteral feeding: a randomized prospective comparison with standard enteral and low calorie/low fat i.v. solutions. Nutrition. 1996 Jun;12(6):423-9. doi: 10.1016/s0899-9007(96)00096-2. PMID 8875537
- [Background] Senkal M, Mumme A, Eickhoff U, Geier B, Spath G, Wulfert D, Joosten U, Frei A, Kemen M. Early postoperative enteral immunonutrition: clinical outcome and cost-comparison analysis in surgical patients. Crit Care Med. 1997 Sep;25(9):1489-96. doi: 10.1097/00003246-199709000-00015. PMID 9295822
- [Background] Tsekos E, Reuter C, Stehle P, Boeden G. Perioperative administration of parenteral fish oil supplements in a routine clinical setting improves patient outcome after major abdominal surgery. Clin Nutr. 2004 Jun;23(3):325-30. doi: 10.1016/j.clnu.2003.07.008. PMID 15158295
- [Background] Weiss G, Meyer F, Matthies B, Pross M, Koenig W, Lippert H. Immunomodulation by perioperative administration of n-3 fatty acids. Br J Nutr. 2002 Jan;87 Suppl 1:S89-94. doi: 10.1079/bjn2001461. PMID 11895158
- [Background] Wachtler P, Konig W, Senkal M, Kemen M, Koller M. Influence of a total parenteral nutrition enriched with omega-3 fatty acids on leukotriene synthesis of peripheral leukocytes and systemic cytokine levels in patients with major surgery. J Trauma. 1997 Feb;42(2):191-8. doi: 10.1097/00005373-199702000-00004. PMID 9042869
- [Background] Braga M, Vignali A, Gianotti L, Cestari A, Profili M, Di Carlo V. Benefits of early postoperative enteral feeding in cancer patients. Infusionsther Transfusionsmed. 1995 Oct;22(5):280-4. doi: 10.1159/000223143. PMID 8924741
- [Background] Di Carlo V, Gianotti L, Balzano G, Zerbi A, Braga M. Complications of pancreatic surgery and the role of perioperative nutrition. Dig Surg. 1999;16(4):320-6. doi: 10.1159/000018742. PMID 10449977
- [Background] Heslin MJ, Latkany L, Leung D, Brooks AD, Hochwald SN, Pisters PW, Shike M, Brennan MF. A prospective, randomized trial of early enteral feeding after resection of upper gastrointestinal malignancy. Ann Surg. 1997 Oct;226(4):567-77; discussion 577-80. doi: 10.1097/00000658-199710000-00016. PMID 9351723
- [Background] McCarter MD, Gentilini OD, Gomez ME, Daly JM. Preoperative oral supplement with immunonutrients in cancer patients. JPEN J Parenter Enteral Nutr. 1998 Jul-Aug;22(4):206-11. doi: 10.1177/0148607198022004206. PMID 9661120
- [Background] Beier-Holgersen R, Boesby S. Influence of postoperative enteral nutrition on postsurgical infections. Gut. 1996 Dec;39(6):833-5. doi: 10.1136/gut.39.6.833. PMID 9038665
- [Background] Beier-Holgersen R, Brandstrup B. Influence of early postoperative enteral nutrition versus placebo on cell-mediated immunity, as measured with the Multitest CMI. Scand J Gastroenterol. 1999 Jan;34(1):98-102. doi: 10.1080/00365529950172907. PMID 10048740
- [Background] Meydani SN. Effect of (n-3) polyunsaturated fatty acids on cytokine production and their biologic function. Nutrition. 1996 Jan;12(1 Suppl):S8-14. PMID 8850212
- [Background] Brandstrup B, Tonnesen H, Beier-Holgersen R, Hjortso E, Ording H, Lindorff-Larsen K, Rasmussen MS, Lanng C, Wallin L, Iversen LH, Gramkow CS, Okholm M, Blemmer T, Svendsen PE, Rottensten HH, Thage B, Riis J, Jeppesen IS, Teilum D, Christensen AM, Graungaard B, Pott F; Danish Study Group on Perioperative Fluid Therapy. Effects of intravenous fluid restriction on postoperative complications: comparison of two perioperative fluid regimens: a randomized assessor-blinded multicenter trial. Ann Surg. 2003 Nov;238(5):641-8. doi: 10.1097/01.sla.0000094387.50865.23. PMID 14578723
- [Background] Raitt MH, Connor WE, Morris C, Kron J, Halperin B, Chugh SS, McClelland J, Cook J, MacMurdy K, Swenson R, Connor SL, Gerhard G, Kraemer DF, Oseran D, Marchant C, Calhoun D, Shnider R, McAnulty J. Fish oil supplementation and risk of ventricular tachycardia and ventricular fibrillation in patients with implantable defibrillators: a randomized controlled trial. JAMA. 2005 Jun 15;293(23):2884-91. doi: 10.1001/jama.293.23.2884. PMID 15956633
- [Background] Wu D, Meydani SN. n-3 polyunsaturated fatty acids and immune function. Proc Nutr Soc. 1998 Nov;57(4):503-9. doi: 10.1079/pns19980074. PMID 10096109
- [Derived] Sorensen LS, Thorlacius-Ussing O, Schmidt EB, Rasmussen HH, Lundbye-Christensen S, Calder PC, Lindorff-Larsen K. Randomized clinical trial of perioperative omega-3 fatty acid supplements in elective colorectal cancer surgery. Br J Surg. 2014 Jan;101(2):33-42. doi: 10.1002/bjs.9361. Epub 2013 Nov 26. PMID 24281905
- [Derived] Sorensen LS, Rasmussen HH, Aardestrup IV, Thorlacius-Ussing O, Lindorff-Larsen K, Schmidt EB, Calder PC. Rapid incorporation of omega-3 fatty acids into colonic tissue after oral supplementation in patients with colorectal cancer: a randomized, placebo-controlled intervention trial. JPEN J Parenter Enteral Nutr. 2014 Jul;38(5):617-24. doi: 10.1177/0148607113491782. Epub 2013 Jun 20. PMID 23788002